CLINICAL TRIAL: NCT03313739
Title: The Effect of an Educational Intervention Based on the Teach Back Method on Self-care Practice Among Menopausal Women
Brief Title: An Educational Intervention Based on the Teach Back Method on Self-care Practice Among Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonabad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Narjes Bahri, Dr. Narjes Bahri, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P/4/69
Record Dates: First submitted 2017-10-11; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An Educational Program
  Interventions: Other: An Educational Program
- Control group (No Intervention): This group(n=30) received no intervention.

INTERVENTIONS:
Other: An Educational Program — An educational program was designed for self-care during menopause using teach back method.
  Arms: Intervention group

SUMMARY:
This study was conducted to assess the effects of an educational program that had designed based on teach back method in order to improve self-care competency among menopausal women.

DETAILED DESCRIPTION:
In this study 60 menopausal women randomly allocated to intervention group(n=30) and control group(n=30).

Intervention group participated in an educational program that had designed in four sessions based on teach back method. Control group revived no education.

ELIGIBILITY:
Inclusion Criteria:

* menopausal women(1-5 years after menopause)
* no history of hysterectomy
* no history of oophorectomy
* literacy for reading and writing

Exclusion Criteria:

* no interest for continuing the study
* no participating in all educational sessions

Ages: 46 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
self-care practice | one month
  self-care practice regard menopausal health was measured using a researcher made questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Narjes Bahri, PhD, Study Director — GMU

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bahri N, Yoshany N, Morowatisharifabad MA, Noghabi AD, Sajjadi M. The effects of menopausal health training for spouses on women's quality of life during menopause transitional period. Menopause. 2016 Feb;23(2):183-8. doi: 10.1097/GME.0000000000000588. PMID 26783984
- See also: related paper — https://www.ncbi.nlm.nih.gov/pubmed/26783984